CLINICAL TRIAL: NCT02121392
Title: Continuous Adductor Canal Block With Epidural Analgesia for Total Knee Arthroplasty: A Prospective, Randomized, Double-blinded, Placebo-Controlled Trial
Brief Title: Epidural Catheter With or Without Adductor Canal Nerve Block for Postoperative Analgesia Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB13-1438
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Arthroplasty, Replacement, Knee; Nerve Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural Catheter without Adductor Canal Nerve Block Catheter (Sham Comparator): Patients randomized to the sham catheter will have a sham catheter placed on the skin and obscured with an opaque dressing and attached to a functional pump which will not be turned on.
  Interventions: Device: Adductor Canal Nerve Block Sham Catheter; Drug: Bupivacaine
- Epidural Catheter with Adductor Canal Nerve Block Catheter (Experimental): Patients will receive a continuous adductor canal block placed under ultrasound guidance under the supervision of an attending physician who is fellowship trained.
  Interventions: Device: Adductor Canal Nerve Block Catheter; Drug: Bupivacaine

INTERVENTIONS:
Device: Adductor Canal Nerve Block Catheter — ACNB catheter will be placed by anesthesia residents under the supervision of board-certified anesthesiologists familiar with regional anesthesia techniques, who are part of the anesthesia pain service. They will be performed at the bedside, aseptically, with the patient's vital signs monitored throughout the procedure. 1% lidocaine will be infiltrated in the skin and subcutaneous tissues overlying the adductor canal as visualized on ultrasound. Via a 17 gauge touhy needle a closed tip non-stimulating, epidural catheter will be placed after 1% lidocaine is used to hydrodissect the space lateral to the superficial femoral artery within the adductor canal. The catheter will be secured to the skin. All catheters will be connected to infusion pumps with opaque plastic bags covering the pumps. The functional ACNB pumps will run 8cc/h.
  Arms: Epidural Catheter with Adductor Canal Nerve Block Catheter
Device: Adductor Canal Nerve Block Sham Catheter — Patients randomized to the sham catheter will have a chlorhexidine prep of the skin and ultrasound examination of the adductor canal on postoperative day #1. To minimize patient risk, a wooden applicator will be used to apply 10 seconds of pressure to the leg followed by catheter securing to the skin with the same tegaderm and paper tape dressing used on functional catheters. All catheters will be connected to infusion pumps with opaque plastic bags covering the pumps. The sham catheter pumps will not be turned on.
  Arms: Epidural Catheter without Adductor Canal Nerve Block Catheter
Drug: Bupivacaine — In the functioning continuous adductor canal block, 0.125% bupivacaine will be infused at a rate of 8cc/hr.

SUMMARY:
The purpose of this study is to further investigate the efficacy of adductor canal nerve blocks for pain management after total knee replacement. Specifically we are studying adductor canal nerve blocks in conjunction with epidural anesthesia, which is a combination that has not been extensively researched before. Our question is whether combining these modalities will enhance patient satisfaction after surgery and accelerate patients' readiness to discharge.

DETAILED DESCRIPTION:
Knee replacement surgery has become increasingly more common in the United States with hundreds of thousands of surgeries performed yearly across the country. Despite that, there is no consensus "standard of care" for optimum pain control regimen after surgery. Pain management after TKA ranges from local tissue injections and patient controlled anesthesia to regional nerve blocks to neuraxial anesthesia. Although regional anesthesia has become more common and widespread, there are wide variations depending on practice setting (academic versus private), equipment available (adductor nerve blocks require ultrasound guidance), level of training of the anesthesiologists and patient selection, among other factors. Another part of the reason for the wide variations in practice is the lack of literature demonstrating clear effectiveness or superiority of one technique over another.

To date adductor canal nerve blocks have been mainly studied in comparison with femoral nerve blocks in terms of their efficacy in controlling pain and their ability to preserve motor function. Adductor canal nerve blocks have been shown in the literature to be an effective method for postoperative pain control in total knee replacement surgery. One of the unique benefits of this particular technique is that the adductor canal nerve block is primarily a sensory block, thereby controlling pain without impairing motor strength. This is useful for total knee replacement surgery as pain is controlled while quadriceps muscle strength is preserved. With well functioning muscles patients are able to fully participate in physical therapy with less strength impairment and reduced risk of falling.

It is our aim to investigate one multimodal approach that combines the strengths of two proven pain management techniques and thereby improve overall postoperative pain control and patient satisfaction. Our hope is to establish a protocol that is safe and effective for patient care.

ELIGIBILITY:
Inclusion Criteria:

* end stage degenerative joint disease
* enrolled for unilateral total knee arthroplasty at the University of Chicago
* age < 85
* ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* age > 85
* American Society of Anesthesiologists physical status > 3
* known hypersensitivity to lidocaine, bupivacaine, ropivacaine or other local anesthetic agents
* Coagulopathy, specifically INR > 1.5, Platelets < 100, therapy with clopidogrel within 5 days prior to surgery, enoxaparin or fondaparinux within the last 24 hours prior to surgery, patients with anti-phospholipid syndrome requiring aggressive anticoagulation perioperatively
* History of alcohol or substance abuse (including strong opioids - morphine, oxycodone, methadone, fentanyl, ketobemidone), taking > 50 mg morphine equivalent daily of opioids
* Pre-existing femoral neuropathy or radiculopathy
* Patients with poor ability to communicate

Max Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hue Luu, MD, Principal Investigator — University of Chicago; Magdalena Anitescu, MD, Principal Investigator — University of Chicago; David Dickerson, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

REFERENCES:
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Grevstad U, Mathiesen O, Lind T, Dahl JB. Effect of adductor canal block on pain in patients with severe pain after total knee arthroplasty: a randomized study with individual patient analysis. Br J Anaesth. 2014 May;112(5):912-9. doi: 10.1093/bja/aet441. Epub 2014 Jan 8. PMID 24401802
- [Background] Mudumbai SC, Kim TE, Howard SK, Workman JJ, Giori N, Woolson S, Ganaway T, King R, Mariano ER. Continuous adductor canal blocks are superior to continuous femoral nerve blocks in promoting early ambulation after TKA. Clin Orthop Relat Res. 2014 May;472(5):1377-83. doi: 10.1007/s11999-013-3197-y. PMID 23897505
- [Background] Henningsen MH, Jaeger P, Hilsted KL, Dahl JB. Prevalence of saphenous nerve injury after adductor-canal-blockade in patients receiving total knee arthroplasty. Acta Anaesthesiol Scand. 2013 Jan;57(1):112-7. doi: 10.1111/j.1399-6576.2012.02792.x. Epub 2012 Oct 17. PMID 23074997
- [Background] Ishiguro S, Yokochi A, Yoshioka K, Asano N, Deguchi A, Iwasaki Y, Sudo A, Maruyama K. Technical communication: anatomy and clinical implications of ultrasound-guided selective femoral nerve block. Anesth Analg. 2012 Dec;115(6):1467-70. doi: 10.1213/ANE.0b013e31826af956. Epub 2012 Aug 10. PMID 22886842
- [Background] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Derived] Leung P, Dickerson DM, Denduluri SK, Mohammed MK, Lu M, Anitescu M, Luu HH. Postoperative continuous adductor canal block for total knee arthroplasty improves pain and functional recovery: A randomized controlled clinical trial. J Clin Anesth. 2018 Sep;49:46-52. doi: 10.1016/j.jclinane.2018.06.004. Epub 2018 Jun 8. PMID 29890381

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Catheter With Adductor Canal Nerve Block Catheter: Patients will receive a continuous adductor canal block placed under ultrasound guidance under the supervision of an attending physician who is fellowship trained.
  Adductor Canal Nerve Block Catheter: ACNB catheter will be placed by anesthesia residents under the supervision of board-certified anesthesiologists familiar with regional anesthesia techniques, who are part of the anesthesia pain service. They will be performed at the bedside, aseptically, with the patient's vital signs monitored throughout the procedure. 1% lidocaine will be infiltrated in the skin and subcutaneous tissues overlying the adductor canal as visualized on ultrasound. Via a 17 gauge touhy needle a closed tip non-stimulating, epidural catheter will be placed after 1% lidocaine is used to hydrodissect the space lateral to the superficial femoral artery within the adductor canal. The catheter will be secured to the skin. All catheters will be connected to infusion pumps with opaque plastic bags covering the
Period: Prior to Intervention
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Started | 83 | 82
Completed | 35 | 41
Not Completed | 48 | 41
Not completed — Protocol Violation | 40 | 35
Not completed — Withdrawal by Subject | 8 | 6
Period: After Placement of AC Block vs Sham
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Started | 35 | 41
Completed | 32 | 38
Not Completed | 3 | 3
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: In the cACB group, 39 patients were included in the analysis of the inpatient variables. 1 patient was lost to outpatient follow-up and thus there are 38 patient ultimately in the cACB group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter | Total
Number analyzed (Participants) | 32 | 39 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.18 (10.35) | 64.44 (8.77) | 63.87 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 7 | 9 | 16
American Society of Anaesthesiologists Score [Mean (Standard Deviation); unit: units on a scale] — The American Society of Anesthesiologists (ASA) scoring system is a 6-category scale and is widely used to assess patients' general preoperative health:
  1. A normal healthy patient
  2. A patient with mild systemic disease
  3. A patient with severe systemic disease
  4. A patient with severe systemic disease that is a constant threat to life
  5. A moribund patient who is not expected to survive without the operation
  6. A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2.66 (0.48) | 2.79 (0.41) | 2.68 (0.47)
Body Mass Index (Kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 34.38 (6.14) | 33.58 (7.11) | 33.94 (6.65)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) [Mean (Standard Deviation); unit: units on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain (5 items), stiffness (2 items), and physical function (17 items). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores represent worse pain, stiffness, and functional limitations. A sum of the scores for all three subscales yields a total WOMAC score.
  units on a scale | 51.68 (14.23) | 50.78 (18.94) | 51.19 (16.85)
knee extension (deg) [Mean (Standard Deviation); unit: degrees] | 1.54 (3.00) | 4.24 (7.14) | 3.02 (5.78)
knee flexion (deg) [Mean (Standard Deviation); unit: degrees] | 103.43 (18.62) | 97.41 (26.23) | 100.13 (23.12)
knee Range of motion (deg) [Mean (Standard Deviation); unit: degrees] | 101.89 (19.97) | 93.18 (27.24) | 97.11 (24.43)

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalents
Time Frame: 12 hours postoperatively and 20 hours after placement of catheter
Measure: Mean (Standard Deviation); unit: milligrams of morphine
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
milligrams of morphine
  12 hours postoperatively | 11.9 (14) | 12.5 (15)
  20 hours after placement of catheter | 96.5 (47) | 73.9 (38)

2. Secondary Outcome: Visual Analog Score for Pain
Description: The visual analog scale (VAS) is a pain rating scale. Scores are based on self-reported measures of symptoms that are recorded with a single mark placed at one point along the length of a line that represents a continuum between the two ends of the scale-"no pain" on the left end of the scale (equal to a score of 0) and the "worst pain" on the right end of the scale (equal to a score of 100).
Time Frame: 12 hours postoperatively and 20 hours after placement of catheter
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
mm
  12 hours postoperatively | 27.9 (16) | 26.9 (19)
  20 hours after placement of catheter | 36.4 (18) | 28.6 (14)

3. Secondary Outcome: Physical Therapy Ambulation Distance
Time Frame: Daily on postoperative days one and two
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
meters
  Postoperative Day 1 | 13.8 (15.6) | 17.6 (21)
  Postoperative Day 2 | 32.5 (26.2) | 39.4 (31.8)

4. Secondary Outcome: Number of Hospital Days Until Discharge Criteria Are Met
Time Frame: within first 3 days (plus or minus 3 days) after surgery
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
Days | 2.42 (0.86) | 2.67 (1.1)

5. Secondary Outcome: Number of Participants With Bleeding Complications at Adductor Canal Nerve Block Catheter Site
Time Frame: within first 3 days (plus or minus 3 days) after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events Related to Adductor Canal Nerve Block Catheter
Time Frame: within first 3 days (plus or minus 3 days) after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
Participants | 0 | 0

7. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self administered questionnaire consisting of 24 items divided into 3 subscales: pain (5 items), stiffness (2 items), and physical function (17 items). The subscale scores can vary, with pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores represent worse pain, stiffness, and functional limitations. A sum of the scores for all three subscales yields a total WOMAC score.
Time Frame: 3 and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 38
score on a scale
  3 weeks | 37.8 (13) | 29.1 (15)
  6 weeks | 32.9 (14) | 27.9 (17)

8. Secondary Outcome: Range of Motion
Description: Knee range of motion (ROM) was measured (in degrees) during physical therapy.
Time Frame: postoperative day 1 and 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
degrees
  Postoperative Day 1 | 51.4 (17) | 40.6 (14)
  Postoperative Day 2 | 71.3 (19) | 62.5 (21)

9. Secondary Outcome: Range of Motion at 3 and 6 Week Follow up
Time Frame: 3 and 6 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
Number analyzed (Participants) | 32 | 39
degrees
  3 weeks | 98.2 (11.5) | 94.3 (13)
  6 weeks | 109 (14) | 105 (10.2)

ADVERSE EVENTS:
Time Frame: Following placement of catheter until removal immediately prior to discharge, an average of 2.5 days
Description: Adverse Events were recorded only for patients in whom the catheter was successfully placed (i.e., those who progressed to period titled "After Placement of AC Block vs Sham"). There were no adverse events associated with catheter placement.
Arm/Group | Epidural Catheter Without Adductor Canal Nerve Block Catheter | Epidural Catheter With Adductor Canal Nerve Block Catheter
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/41
Other Adverse Events (participants affected / at risk) | 0/35 | 0/41

LIMITATIONS AND CAVEATS:
Limitations included the number of patients withdrawn (n = 89) after randomization. The majority withdrew due to unsuccessful epidural catheterization (n = 34). Despite this, these patients were distributed evenly across the two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes